CLINICAL TRIAL: NCT05550831
Title: Radiofrequency Before to Surgical Removal of a Recalcitrant Morton´s Neuroma
Acronym: REQUIEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Alfonso Martínez Nova, Doctor, Universidad de Extremadura
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REQUIEM
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Morton Neuroma; Radriofrequency
Keywords: Foot; Morton Neuroma; Radiofrequency
MeSH Terms: conditions — Morton Neuroma

STUDY DESIGN:
Intervention Model Description: Performing a radiofrequency procedure prior to the removal of morton's neuroma. This procedure would be performed to check in which percentage of the nerve ablation has been performed, and whether the current protocol is performed correctly or parts of the nerve remain intact.
  * Step 1: Visualize the needle on the long axis of the probe.
  * Step 2: Neurostimulate
  * Step 3: Deposit of 1-2cc of anesthetic and wait about 2 minutes.
  * Step 4: we apply the continuous radiofrequency at that point and once done we change the position of the needle to more dorsal planes anatomically and we made 2 more applications (in this case we will no longer have neurostimulation because the patient will be anesthetized).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency (Experimental): Radiofrequency procedure prior to the removal of morton's neuroma.
  * Radiofrequency Machine: Multilesion Generator 3 Channels TLG-10 STP.
  * Temperature: 80-85ºC
  * Time: 90 seconds
  * Active needle size: 1 cm
  * Number of Applications: 3
  * Impedance: less than 550
  * Ultrasound. General Electric Logic R7 with 12 Mgh probe.
  Interventions: Procedure: Radiofrequency

INTERVENTIONS:
Procedure: Radiofrequency — Peripheral ablation of affected Morton´s Neuroma nerve endings by thermal dissipation by an electrode.

SUMMARY:
The purpose of this study is to perform a radiofrequency procedure prior to the removal of morton's neuroma. This procedure would be performed to check in which percentage of the nerve ablation has been performed, and whether the current protocol is performed correctly or parts of the nerve remain intact.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 70 years
* Patient with neuroma of morton of more than 1 year of evolution
* Patient treated by conservative treatments, stencils, various infiltrations, stretching and with symptomatology that limits his daily activities.
* Healthy patients without previous systemic pathologies (diabetes, coagulation or immunological disorders), ASA I or II that require and demand surgical treatment of their pathology in the participating centers and willing to participate in the study.
* freely accept and sign the informed consent for participation in the study.

Exclusion Criteria:

* Allergy to local anesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Nerve Damage | 1 week
  Anatomopathology of the nerve
Quality of Life, FFI | 6 months
  FFI Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Alfonso Martínez Nova, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: Undecided